CLINICAL TRIAL: NCT04237662
Title: The Impact of Enamel Matrix Derivatives on Periodontal Healing in Diabetic Patients After Non-Surgical Periodontal Therapy
Brief Title: Enamel Matrix Derivatives & Periodontal Therapy in Diabetic Patients
Acronym: PERIOEMD-4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Full Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3649-2019
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Single-centre randomized, parallel design, clinical trial with a 3-month follow-up
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Opaque envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Root Instrumentation + Enamel Matrix Derivative Application
  Periodontal treatment is delivered with ultrasonic instrumentation performed with fine tips. The approach chosen is the one- stage full-mouth ultrasonic debridement in which all the treatment of diseased sites is performed within one hour.
  In this group, at the end of the instrumentation enamel matrix derivatives is placed in all sites with a periodontal pocket depth deeper than 5mm.
  Interventions: Procedure: Root Instrumentation; Device: Enamel Matrix Derivative application
- Control Group (Active Comparator): Root Instrumentation
  Periodontal treatment is delivered with ultrasonic instrumentation performed with fine tips. The approach chosen is the one- stage full-mouth ultrasonic debridement in which all the treatment of diseased sites is performed within one hour.
  Interventions: Procedure: Root Instrumentation

INTERVENTIONS:
Procedure: Root Instrumentation — Instrumentation of the root surface in order to achieve debridement
Device: Enamel Matrix Derivative application — Enamel Matrix Derivative will be applied in the sites with at least 6 mm of pocket depths
  Arms: Test Group

SUMMARY:
The aim of this study is to compare periodontal treatment with or without the adjunct of an enamel matrix derivative in terms of periodontal healing in diabetic patients.

DETAILED DESCRIPTION:
Patients with periodontitis will be randomly allocated to two groups. In both groups, periodontal root instrumentation will be performed. In the test group, an additional flapless application of enamel matrix derivatives will be granted for sites with pockets deeper than 5 mm.

Metabolic glucose control as measured through blood testing and local parameters of periodontal health will be measured at baseline and three months after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diabetes mellitus type II and currently under treatment;
* No previous periodontal treatment in the last 6 months;
* Presence of Periodontitis (Clinical attachment loss of at least 3 mm in 2 or more non- adjacent teeth);
* Ability to understand the study procedures and comply with them through the length of the study.

Exclusion Criteria:

* Pregnancy and breast feeding;
* Need for antibiotic treatment during periodontal therapy;
* Chronic infections;
* Systemic diseases;
* Patients who report current smoking over 20 cigarettes per day.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pocket probing depth (PPD) | Measured at Baseline and 3 months after treatment
  Changes in PPD, measured orally through clinical examination. Unit of measure: mm

SECONDARY OUTCOMES:
Clinical attachment level (CAL) | Measured at Baseline and 3 months after treatment
  Changes in CAL, measured orally through clinical examination. Unit of measure: mm
Recession of the gingival margin (REC) | Measured at Baseline and 3 months after treatment
  Changes in REC, measured orally through clinical examination. Unit of measure: mm
Number of sites with Pocket probing depth deeper than 5mm | Measured at Baseline and 3 months after treatment
  Changes, measured orally through clinical examination. Unit of measure: N
Percentage of sites with Pocket probing depth deeper than 5mm | Measured at Baseline and 3 months after treatment
  Changes, measured orally through clinical examination. Unit of measure: %
Percentage of bleeding sites which measured Pocket probing depth deeper than 5mm at baseline | Measured at Baseline and 3 months after treatment
  Changes, measured orally through clinical examination. Unit of measure: %
Full-mouth plaque score (FMPS) | Measured at Baseline and 3 months after treatment
  Changes in Full-mouth plaque score, measuring the amount of dental plaque on the teeth orally through clinical examination. Unit of measure %. The scale ranges from 0% (minimum value, i.e. plaque absent) to 100% (maximum value: all areas are occupied by plaque). 0% would the ideal value. No sub-scales are included.
Full-mouth bleeding score (FMBS) | Measured at Baseline and 3 months after treatment
  Changes of Full-mouth bleeding score, measuring the number of gingival areas that bleed after gingival probe passage. It is measured oral through clinical examination. Unit of measure %. The scale ranges from 0% (minimum value, i. e. gingival inflammation is absent) to 100% (maximum value: all gingival areas are inflamed). 0% would be the ideal value. No sub-scales are included.
Oral Health Index Profile-14 (OHIP-14) | Measured at Baseline and 3 months after treatment
  Changes in Oral Health Index Profile-14 measured through administration of specific questionnaire . Responses for the questionnaire are made on a Likert-type five-point scale, coded 0 (never), 1 (hardly ever), 2 (occasionally), 3 (fairly often), and 4 (very often); with scores ranging from 0-56 and higher scores indicating worse
Oxford Happiness Questionnaire (OHQ) | Measured at Baseline and 3 months after treatment
  Responses for the questionnaire are made on a Likert scale, coded from strongly disagree = 1 to strongly agree = 6, with the higher scores corresponding to higher levels of happiness. For the 12 negatively worded items, the reverse coding is necessary before calculating the total score, which is a sum of individual item scores. Score range is from 1 as a minimum and 6 as a maximum score.
High sensitivity C-Reactive Protein (hsCRP) | Measured at Baseline and 3 months after treatment
  analyzed through blood sampling. Unit of measure: mg/L
Glycated Hemoglobin (HbA1c) | Measured at Baseline and 3 months after treatment
  analyzed through blood sampling. Unit of measure: mmol/mol

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graziani F, Gennai S, Petrini M, Bettini L, Tonetti M. Enamel matrix derivative stabilizes blood clot and improves clinical healing in deep pockets after flapless periodontal therapy: A Randomized Clinical Trial. J Clin Periodontol. 2019 Feb;46(2):231-240. doi: 10.1111/jcpe.13074. PMID 30663788